CLINICAL TRIAL: NCT01091194
Title: Effect of High Intensity Interval-based Aerobic Exercise 1-8 Years After Heart Transplantation. 1 Year Follow Up.
Brief Title: Effect of Exercise After Heart Transplantation
Acronym: TEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10920
Record Dates: First submitted 2010-03-18; First posted 2010-03-23 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Heart Transplantation
Keywords: Heart Transplantation; Aerobic Exercise; Exercise, Physical; Exercise Test; Treadmill Test; VO2 peak; Muscle Strength; Quality of Life; Reinnervation; Heart Rate; Myocardial Function
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Other): Interval-based aerobic exercise
  Interventions: Other: Interval-based aerobic exercise
- Control (No Intervention): No intervention other than regular follow up hospital visits

INTERVENTIONS:
Other: Interval-based aerobic exercise — High intensity interval-based aerobic exercise training. Duration: 1 year. Three 8-weeks supervised periods of physical training 3 times per week. Individual training 2 times per week between these periods.
  Other Names: physical activity, fitness
  Arms: Exercise

SUMMARY:
This is a randomized controlled trial which will include approximately 50 heart transplant recipients 1-8 years after heart transplantation. The intervention and follow up period is 1 year. The primary purpose is to investigate if systematic, high intensity, interval-based aerobic exercise training results in a greater improvement of exercise capacity (measured by VO2peak) than previously shown in heart transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Norwegian heart transplanted patients > 18 years of age
* 1-8 years after heart transplantation
* Optimal medical treatment
* Stable condition
* Written informed consent
* Must have access to a physical therapist or personal trainer in their hometown
* Motivation for exercise

Exclusion Criteria:

* Unstable condition
* In need of revascularization or other invention
* Infections, open wounds or skin diseases
* Physical disabilities which prevent participation
* Other diseases, illnesses or conditions which contradict exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2peak) | Before and after the intervention period of 1 year

SECONDARY OUTCOMES:
Isokinetic muscle strength of quadriceps and hamstrings | Before and after the intervention period of 1 year
Quality of life measured by questionnaires | Before and after the intervention period of 1 year
Myocardial function measured by echocardiography | Before and after the intervention period of 1 year
Progression on coronary atherosclerosis measured by intra vascular ultrasound (IVUS) | Before and after the intervention period of 1 year
Vascular tone and compliance measured by tonometry | Before and after the intervention period of 1 year
Regular blood screening, lipid profile, inflammatory status, nerve growth factor, biochemical markers for endothelial function, prothrombotic factor, factors connected to vascularization: NT-proBNP and gene expression analysis. | Before and after the intervention period of 1 year
Analysis of isolated muscle cells from myocardial biopsy | Before and after the intervention period of 1 year
Reinnervation as judged by autonomic nervous control (Heart Rate Variability) | Before and after the intervention period of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, MD,PhD,Prof., Study Director — Oslo University Hospital
Locations (1):
- Department of Cardiology, Oslo University Hospital, Rikshospitalet, Oslo, Norway

REFERENCES:
- [Result] Nytroen K, Rustad LA, Aukrust P, Ueland T, Hallen J, Holm I, Rolid K, Lekva T, Fiane AE, Amlie JP, Aakhus S, Gullestad L. High-intensity interval training improves peak oxygen uptake and muscular exercise capacity in heart transplant recipients. Am J Transplant. 2012 Nov;12(11):3134-42. doi: 10.1111/j.1600-6143.2012.04221.x. Epub 2012 Aug 17. PMID 22900793
- [Result] Rustad LA, Nytroen K, Amundsen BH, Gullestad L, Aakhus S. One year of high-intensity interval training improves exercise capacity, but not left ventricular function in stable heart transplant recipients: a randomised controlled trial. Eur J Prev Cardiol. 2014 Feb;21(2):181-91. doi: 10.1177/2047487312469477. Epub 2012 Nov 26. PMID 23185084
- [Result] Nytroen K, Rustad LA, Gude E, Hallen J, Fiane AE, Rolid K, Holm I, Aakhus S, Gullestad L. Muscular exercise capacity and body fat predict VO(2peak) in heart transplant recipients. Eur J Prev Cardiol. 2014 Jan;21(1):21-9. doi: 10.1177/2047487312450540. Epub 2012 Jun 1. PMID 22659939
- [Derived] Nytroen K, Rolid K, Yardley M, Gullestad L. Effect of high-intensity interval training in young heart transplant recipients: results from two randomized controlled trials. BMC Sports Sci Med Rehabil. 2020 Jun 4;12:35. doi: 10.1186/s13102-020-00180-1. eCollection 2020. PMID 32518655